CLINICAL TRIAL: NCT03493945
Title: A Phase I/II Study of Immunotherapy Combination BN-Brachyury Vaccine, M7824, N-803 and Epacadostat (QuEST1)
Brief Title: Phase I/II Study of Immunotherapy Combination BN-Brachyury Vaccine, M7824, N-803 and Epacadostat (QuEST1)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, James Gulley, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 180078; 18-C-0078
Record Dates: First submitted 2018-04-10; First posted 2018-04-11 (Actual); Results first posted 2025-06-08 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Castration-resistant Prostate Cancer; Prostate Cancer; Prostate Neoplasm; Advanced Solid Tumor; Solid Tumor; Non-metastatic Castration-resistant Prostate Cancer
Keywords: Immunotherapy; Combined Treatment; PD-1/PD-L1; Tumor-Specific T Cells; Novel Cancer Vaccine
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bintrafusp alfa protein, human; ALT-803; epacadostat; Acetaminophen; Ibuprofen; Naproxen; Diphenhydramine; Electrocardiography; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Arm 1.1 Bintrafusp alfa (M7824) + Anktiva (N-803) (Experimental): Bintrafusp alfa (M7824) + Anktiva (N-803)
  Interventions: Biological: M7824; Drug: N-803; Drug: Acetaminophen; Drug: Ibuprofen; Drug: Naproxen; Other: Benadryl; Diagnostic Test: EKG; Diagnostic Test: Bone scan; Diagnostic Test: CT chest, abdomen and pelvis; Diagnostic Test: MRI
- Arm 2.1A Bintrafusp alfa (M7824) + Bavarian Nordic (BN)-Brachyury during phase IIA (Experimental): Bintrafusp alfa (M7824) + Bavarian Nordic (BN)-Brachyury during phase IIA
  Interventions: Biological: M7824; Biological: MVA-BN-Brachyury; Biological: FPV-Brachyury; Drug: Acetaminophen; Drug: Ibuprofen; Drug: Naproxen; Other: Benadryl; Diagnostic Test: EKG; Diagnostic Test: Bone scan; Diagnostic Test: CT chest, abdomen and pelvis; Diagnostic Test: MRI
- Arm 2.1B Bintrafusp alfa (M7824) + Bavarian Nordic (BN)-Brachyury during phase IIB (Experimental): Bintrafusp alfa (M7824) + Bavarian Nordic (BN)-Brachyury during phase IIB
  Interventions: Biological: M7824; Biological: MVA-BN-Brachyury; Biological: FPV-Brachyury; Drug: Acetaminophen; Drug: Ibuprofen; Drug: Naproxen; Other: Benadryl; Diagnostic Test: EKG; Diagnostic Test: Bone scan; Diagnostic Test: CT chest, abdomen and pelvis; Diagnostic Test: MRI
- Arm 2.2A Bintrafusp alfa (M7824) + Bavarian Nordic (BN)-Brachyury + Anktiva (N-803) during phase IIA (Experimental): Bintrafusp alfa (M7824) + Bavarian Nordic (BN)-Brachyury + Anktiva (N-803) during phase IIA
  Interventions: Biological: M7824; Drug: N-803; Biological: MVA-BN-Brachyury; Biological: FPV-Brachyury; Drug: Acetaminophen; Drug: Ibuprofen; Drug: Naproxen; Other: Benadryl; Diagnostic Test: EKG; Diagnostic Test: Bone scan; Diagnostic Test: CT chest, abdomen and pelvis; Diagnostic Test: MRI
- Arm 2.2B Bintrafusp alfa (M7824) + Bavarian Nordic (BN)-Brachyury + Anktiva (N-803) during phase IIB (Experimental): Bintrafusp alfa (M7824) + Bavarian Nordic (BN)-Brachyury + Anktiva (N-803) during phase IIB
  Interventions: Biological: M7824; Drug: N-803; Biological: MVA-BN-Brachyury; Biological: FPV-Brachyury; Drug: Acetaminophen; Drug: Ibuprofen; Drug: Naproxen; Other: Benadryl; Diagnostic Test: EKG; Diagnostic Test: Bone scan; Diagnostic Test: CT chest, abdomen and pelvis; Diagnostic Test: MRI
- Arm 2.3A M7824 + BN-Brachyury + Anktiva (N-803) + Epacadostat during phase IIA (Experimental): Bintrafusp alfa (M7824) + Bavarian Nordic (BN)-Brachyury + Anktiva (N-803) + Epacadostat during phase IIA
  Interventions: Biological: M7824; Drug: N-803; Biological: MVA-BN-Brachyury; Biological: FPV-Brachyury; Drug: Epacadostat; Drug: Acetaminophen; Drug: Ibuprofen; Drug: Naproxen; Other: Benadryl; Diagnostic Test: EKG; Diagnostic Test: Bone scan; Diagnostic Test: CT chest, abdomen and pelvis; Diagnostic Test: MRI
- Arm 2.3B M7824 + BN-Brachyury + Anktiva (N-803) + Epacadostat during phase IIB (Experimental): Bintrafusp alfa (M7824) + Bavarian Nordic (BN)-Brachyury + Anktiva (N-803) + Epacadostat during phase IIB
  Interventions: Biological: M7824; Drug: N-803; Biological: MVA-BN-Brachyury; Biological: FPV-Brachyury; Drug: Epacadostat; Drug: Acetaminophen; Drug: Ibuprofen; Drug: Naproxen; Other: Benadryl; Diagnostic Test: EKG; Diagnostic Test: Bone scan; Diagnostic Test: CT chest, abdomen and pelvis; Diagnostic Test: MRI

INTERVENTIONS:
Biological: M7824 — 1,200 mg intravenous (IV) once every 2 weeks.
  Other Names: Bintrafusp alfa
Drug: N-803 — 8-15 mcg/kg subcutaneous every 2 weeks.
  Other Names: Anktiva
  Arms: Arm 1.1 Bintrafusp alfa (M7824) + Anktiva (N-803); Arm 2.2A Bintrafusp alfa (M7824) + Bavarian Nordic (BN)-Brachyury + Anktiva (N-803) during phase IIA; Arm 2.2B Bintrafusp alfa (M7824) + Bavarian Nordic (BN)-Brachyury + Anktiva (N-803) during phase IIB; Arm 2.3A M7824 + BN-Brachyury + Anktiva (N-803) + Epacadostat during phase IIA; Arm 2.3B M7824 + BN-Brachyury + Anktiva (N-803) + Epacadostat during phase IIB
Biological: MVA-BN-Brachyury — MVA-BN-Brachyury will be administered subcutaneously (2 doses 2 weeks apart).
  Other Names: modified vaccinia Ankara Bavarian Nordic Brachyury
  Arms: Arm 2.1A Bintrafusp alfa (M7824) + Bavarian Nordic (BN)-Brachyury during phase IIA; Arm 2.1B Bintrafusp alfa (M7824) + Bavarian Nordic (BN)-Brachyury during phase IIB; Arm 2.2A Bintrafusp alfa (M7824) + Bavarian Nordic (BN)-Brachyury + Anktiva (N-803) during phase IIA; Arm 2.2B Bintrafusp alfa (M7824) + Bavarian Nordic (BN)-Brachyury + Anktiva (N-803) during phase IIB; Arm 2.3A M7824 + BN-Brachyury + Anktiva (N-803) + Epacadostat during phase IIA; Arm 2.3B M7824 + BN-Brachyury + Anktiva (N-803) + Epacadostat during phase IIB
Biological: FPV-Brachyury — FPV-Brachyury will be given 2 weeks after second dose of modified vaccinia Ankara (MVA)-Bavarian Nordic (BN)-Brachyury, then every 4 weeks until 6 months, then every 3 months for 2 years, then every 6 months.
  Other Names: Fowlpox Virus Brachyury
  Arms: Arm 2.1A Bintrafusp alfa (M7824) + Bavarian Nordic (BN)-Brachyury during phase IIA; Arm 2.1B Bintrafusp alfa (M7824) + Bavarian Nordic (BN)-Brachyury during phase IIB; Arm 2.2A Bintrafusp alfa (M7824) + Bavarian Nordic (BN)-Brachyury + Anktiva (N-803) during phase IIA; Arm 2.2B Bintrafusp alfa (M7824) + Bavarian Nordic (BN)-Brachyury + Anktiva (N-803) during phase IIB; Arm 2.3A M7824 + BN-Brachyury + Anktiva (N-803) + Epacadostat during phase IIA; Arm 2.3B M7824 + BN-Brachyury + Anktiva (N-803) + Epacadostat during phase IIB
Drug: Epacadostat — 600 mg orally twice daily (1200 MG total).
  Other Names: IDO1
  Arms: Arm 2.3A M7824 + BN-Brachyury + Anktiva (N-803) + Epacadostat during phase IIA; Arm 2.3B M7824 + BN-Brachyury + Anktiva (N-803) + Epacadostat during phase IIB
Drug: Acetaminophen — Antipyretic medication, orally, prior to infusion, up to 650mg.
  Other Names: Tylenol; Ofirmev; FeverAll
Drug: Ibuprofen — Antipyretic medication, orally, prior to infusion, up to 600mg.
  Other Names: Advil; Advil Migraine
Drug: Naproxen — Antipyretic medication, orally, prior to infusion, up to 500mg.
  Other Names: Aleve; Naprosyn; Anaprox DS
Other: Benadryl — 50mg orally prior to infusion.
  Other Names: Diphenhydramine
Diagnostic Test: EKG — Baseline and principal investigator discretion.
  Other Names: Electrocardiogram
Diagnostic Test: Bone scan — Restaging every 12 weeks.
  Other Names: Bone scintigraphy
Diagnostic Test: CT chest, abdomen and pelvis — Every 12 weeks after start of therapy.
  Other Names: Computed tomography chest, abdomen and pelvis
Diagnostic Test: MRI — If clinically indicated.
  Other Names: Magnetic resonance imaging

SUMMARY:
Background:

Immunotherapy drugs help the body to fight cancer. Scientists think that combining some of these drugs will make them work better than when used alone. This may be true for many types of cancer, including castration-resistant prostate cancer (CRPC).

Objective:

To test if any of the combinations of drugs below have anti-prostate cancer activity and to test if they are safe.

1. Bavarian-Nordic (BN)-brachyury, bintrafusp alfa (M7824).
2. Bavarian-Nordic (BN)-brachyury, bintrafusp alfa (M7824) + Anktiva (N-803).
3. Bavarian-Nordic (BN)-brachyury, bintrafusp alfa (M7824) + Anktiva (N-803) + Epacadostat.

Eligibility:

People ages 18 and older with CRPC or another metastatic cancer

Design:

Participants will be screened with:

* Medical history
* Physical exam
* Computed tomography (CT) or magnetic resonance imaging (MRI) scans
* Possible bone imaging
* Blood, urine, and heart tests
* Possible tumor biopsy

Participants will be treated with a 2-, 3- or 4-drug combinations of the following study drugs in 2-week cycles:

* Participants will receive M7824 by intravenous (IV) once every 2 weeks.
* Participants will receive N-803 by injection once every 2 weeks. They will record any skin changes at the injection site in a diary.
* Participants will receive BN-brachyury as 4 injections to different limbs. They will get the first 3 doses 2 weeks apart. Then they will get doses every 4 weeks for 6 months, then every 3 months for 2 years, then every 6 months.
* Participants will take Epacadostat orally every 12 hours. They will keep a pill diary.

Participants will have physical exams and blood and urine tests at the start of each cycle. They may have scans every 12 weeks.

Participants will continue treatment until their disease gets worse or they cannot tolerate the side effects.

Participants will have a follow-up visit 4-5 weeks after they stop treatment. They will have a physical exam and blood tests. They may be asked to return for scans every 3 months.

DETAILED DESCRIPTION:
Background:

* Programmed cell death protein 1 (PD-1)/programmed death ligand 1 (PD-L1) signaling appears to be a major inhibitor of activated T cell anti-tumor immune responses. The rapid, deep and durable responses seen in various malignancies with PD-1/PD-L1 targeted agents demonstrate that blockade of this axis is key to facilitating immune responses within the tumor microenvironment (TME).
* Prostate cancer is poorly recognized by T cells. Lack of an immune response is one explanation for the lower response rates (<15%) observed with anti-PD-1/PD-L1 therapies for prostate cancer.
* Increasing response rates will likely require therapeutic nullification of multiple immune deficits by combining immunotherapies that generate tumor-specific T cells (vaccine), dampen the inhibitory milieu of the TME, and enhance T and natural killer (NK) cell activity within the TME.
* A quick efficacy seeking trial, utilizing sequential arms offers a means to identify signals of activity for combinations of immunotherapy, added sequentially, in castration resistant prostate cancer (CRPC) participants.
* Bavarian Nordic (BN)-Brachyury is a novel recombinant vector-based therapeutic cancer vaccine designed to induce an enhanced immune response against brachyury, which is overexpressed in many solid tumor types, including prostate adenocarcinoma. BN-Brachyury collectively refers to the priming doses (modified vaccinia Ankara (MVA)-BN-Brachyury) and the boost doses (fowlpox virus (FPV)-Brachyury) of the vaccine platform.
* bintrafusp alfa (M7824) is a bifunctional fusion protein consisting of an anti-programmed death ligand 1 (PD-L1) antibody and the extracellular domain of transforming growth factor beta (TGF- beta) receptor type 2, a TGF-beta trap. M7824 can also mediate antibody-dependent cellular cytotoxicity in vitro.
* Anktiva (N-803) is an interleukin 15 (IL-15)/IL-15R alpha superagonist complex that can enhance NK cell mediated antibody-dependent cell-mediated cytotoxicity (ADCC) and T-cell cytotoxicity.
* Synergistic anti-tumor effects have been observed in vitro when combining M7824 and N-803, and in vivo when combining these agents with tumor vaccine in animal models.
* Indoleamine 2,3-dioxygenase 1 (IDO1) is overexpressed in many solid tumors and can contribute to immune escape by tumor cells. INCB024360 (Epacadostat) is an IDO1 inhibitor under investigation in combination with different immunotherapies in treatment of various malignancies.
* In treating of CRPC, we hypothesize that these agents and their effects will be complementary. Tumor-specific T cells generated by vaccine may become more functional in a TME following treatment with M7824 and Epacadostat. N-803 can further enhance the activity of antigen-specific T cells as well as NK cells.

Objective:

-To determine if there is clinical benefit to any of a set of 3 possible treatments for participants with CRPC:

* BN-Brachyury + M7824
* BN-Brachyury + M7824 + N-803
* BN-Brachyury + M7824 + N-803 + Epacadostat

Eligibility:

* Adults with histologically proven CRPC, or metastatic solid tumor of any type for which there is no standard treatment or standard treatment has failed.
* Adequate organ function as defined by liver, kidney, and hematologic laboratory testing.
* Participants with acquired immune defects, active systemic autoimmune disease, history of organ transplant, history of chronic infections, or history of active inflammatory bowel disease are excluded.

Design:

Open label Phase I/II trial with following randomization during the expansion.

Phase I: Cohort 1, Arm 1.1

-Up to 18 participants with any solid tumor will be enrolled in dose escalation Cohort 1 for treatment in Arm 1.1 (flat dose of M7824 + different dose levels of N-803).

Phase IIA: expansion with sequential enrollment into Cohort 2A, Arms 2.1A, 2.2A and 2.3 A

* Concurrently with the enrollment to Arm 1.1, 13 participants with CRPC will start enrollment in Cohort 2A for treatment in Arm 2.1A (M7824 + BN-Brachyury).
* When safe dosing of N-803 is identified during Phase I, 13 participants have enrolled in arm 2.1A and the first 6 participants, treated in Arm 2.1A, have met safety requirements, 13 participants with CRPC will start enrollment in Cohort 2A for treatment in Arm 2.2A (M7824 + BN-Brachyury + N-803).
* When 13 participants have enrolled in Arm 2.2A and the first 6 participants, treated in Arm 2.2A, have met safety requirements, 13 participants with CRPC will start enrollment in Cohort 2A for treatment in Arm 2.3A (M7824 + BN-Brachyury + N-803 + Epacadostat).

Phase IIB: expansion with randomized enrollment into Cohorts 2D and 2R, Arms 2.1B, 2.2B. and 2.3B

* Each Arm in Cohorts 2D and 2R: 2.1B, 2.2B and 2.3B will be open for additional enrollment (25 evaluable participants total) when the initial 13 participants have accrued, safety requirements are meet and a positive signal (defined as Objective Response by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or sustained prostate-specific antigen (PSA) decrease >= 30% sustained for > 21 days) in >= 2 participants is shown.
* If only one arm is open for additional enrollment, participants will be directly assigned to this arm. If 2 arms are open for additional enrollment, participants will be randomized between these 2 open arms. If 3 arms are open for additional enrollment, participants will be randomized among these 3 open arms.

If there are >= 6 of 25 participants with a positive signal of activity in any expansion arm, that arm will be considered of interest for future studies.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants must have histologically or cytologically confirmed any solid tumor (Cohort 1) or castration-resistant prostate cancer (CRPC), Cohorts 2A, 2D and 2R).

For the Cohort 1, eligible participants must have a histologically, cytologically or radiographically proven metastatic or locally advanced solid tumor of any type, for which there is no curative standard therapy or standard therapy has failed.

Castrate testosterone level (less than 50ng/dl or 1.7nmol/L). (Participants with a malignancy other than prostate cancer are excluded from this criterion).

Radiological confirmation of metastatic disease, or

Progressive disease at study entry defined as one or more of the following criteria occurring in the setting of castrate levels of testosterone:

--Radiographic progression defined as any new or enlarging bone lesions or growing lymph node disease, consistent with prostate cancer

OR

--prostate-specific antigen (PSA) progression defined by sequence of rising values separated by greater than 1 week (2 separate increasing values over a minimum of 1 ng/ml (Prostate Cancer Clinical Trials Working Group 3 (PCWG3) PSA eligibility criteria). If participants had been on flutamide, PSA progression is documented 4 weeks or more after withdrawal. For participants on bicalutamide or nilutamide disease progression is documented 6 or more weeks after withdrawal. The requirement for a 4-6 week withdrawal period following discontinuation of flutamide, nilutamide or bicalutamide only applies to participants who have been on these drugs for at least the prior 6 months. For all other participants they must stop bicalutamide, nilutamide or flutamide the day prior to enrollment.

Asymptomatic or mildly symptomatic form prostate cancer; no use of regularly scheduled opiate analgesics for prostate cancer-related pain. (Participants with a malignancy other than prostate cancer are excluded from this criterion).

Participants must agree to continuation of androgen deprivation therapy (ADT) with a gonadotropin-releasing hormone analogue/antagonist or bilateral orchiectomy. (Participants with a malignancy other than prostate cancer are excluded from this criterion). Participants may also continue oral androgen receptor antagonist/anti-androgen therapy (e.g. enzalutamide or abiraterone) unless enrolling to Arm 2.3A or 2.3B due to concerns regarding Cytochrome P450 (CYP)mediated drug-drug interactions epacadostat.

Participants must have had the following prior therapy:

Testosterone lowering therapy for castration-resistant prostate cancer (CRPC)

In addition to continuation of androgen deprivation therapy (ADT) (unless status post bilateral orchiectomy) eligible patients must have received and had PSA or radiographic progression on enzalutamide (or other oral androgen receptor antagonist e.g. darolutamide or apalutamdide) or abiraterone acetate.

Participants who have tumors known to be microsatellite instability high/mismatch repair deficient or tumor mutational burden high must have received prior pembrolizumab.

Participants with known pathogenic homologous recombination repair mutations for which there is evidence of benefit with poly (adenosine diphosphate-ribose) polymerase (PARP) inhibitors (e.g. BReast CAncer gene 1 (BRCA1). BReast CAncer gene 2 (BRCA2), ataxia-telangiectasia mutated (ATM) must have received prior PARP inhibitor.

Age greater than or equal to 18 years.

Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 1

Participants must have adequate organ and marrow function as defined below:

* Absolute neutrophil count greater than or equal to 1000/mcL
* Platelets greater than or equal to 100,000/mcL
* Hemoglobin greater than or equal to 9.0 g/dL
* Total bilirubin within normal institutional limits; in participants with Gilbert's, less than or equal to 3.0 mg/dL
* Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT) serum glutamic-pyruvic transaminase (SGPT) less than or equal to 2.5X upper limit of normal. For subjects with liver involvement in their tumor, AST less than or equal to 3.5. X upper limit of normal (ULN), ALT less than or equal to 3.5 X ULN, and bilirubin less than or equal to 3.0 is acceptable
* Creatinine within 1.5X upper limit of normal institutional limits

The effects of Bavarian Nordic (BN)-Brachyury, bintrafusp alfa (M7824), Anktiva (N-803), and Epacadostat on the developing human fetus are unknown. For this reason, men and women must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, during the study and maintain such contraception until 4 months following the last dose of any study agent. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her partner s treating physician immediately.

Ability of subject to understand and the willingness to sign a written informed consent document.

Participants with successfully treated hepatitis C virus (HCV) are eligible if HCV viral load is undetectable.

EXCLUSION CRITERIA:

Participants who are immunocompromised as follows:

* Human immunodeficiency virus positivity due to the potential for decreased tolerance, and potential to be at risk for severe side effects with immunotherapies. These concerns are relevant to all drugs, as drug-drug interactions among antiretrovirals and immunotherapies are yet uncharacterized.
* Chronic administration (defined as daily or every other day for continued use greater than 14 days) of systemic corticosteroids or other immune suppressive drugs, within 28 days before treatment on study. Nasal, or inhaled steroid, topical steroid creams and eye drops for small body areas are allowed. Physiologic doses of steroids are permitted, e.g., a participant taking hydrocortisone for adrenal insufficiency or a patient recently on abiraterone (administered with 10 mg of prednisone daily) who is tapering off of prednisone is allowed to continue that taper.
* Participants who have undergone allogeneic peripheral stem cell transplantation, or solid organ transplantation requiring immunosuppression

  * Active autoimmune disease, except participants with type 1 diabetes mellitus, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring current immunosuppression, or with other endocrine disorders on replacement hormones or are not excluded if the condition is well controlled.

Prostate cancer participants with a history of brain/leptomeningeal metastasis, since these participants have a very poor prognosis, and immunotherapy may take time to lead to beneficial clinical effects. Participants with brain or CNS metastases enrolling to arm 1.1 are eligible if they are status post definitive radiotherapy or surgery, and are asymptomatic

History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agents to be used in the cohort the subject will be enrolled into.

Known allergy to eggs, egg products, aminoglycoside antibiotics (for example, gentamicin or tobramycin).

Any condition which, in the opinion of the investigator, would prevent full participation in this trial (including the long-term follow-up), or would interfere with the evaluation of the trial endpoints.

Participants with prior investigational drug, chemotherapy, immunotherapy or any prior radiotherapy (except for palliative bone directed therapy) within the past 28 days prior to enrollment, except if the investigator has assessed that all residual treatment-related toxicities have resolved or are minimal and feel the participant is otherwise suitable for enrollment.

Uncontrolled intercurrent acute or chronic illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (>New York Heart Association Class I), hepatic disease, unstable angina pectoris, serious cardiac arrhythmia, requiring medication, uncontrolled hypertension (Systolic blood pressure (SBP) >170/ diastolic blood pressure (DBP)>105) or psychiatric illness/social situations within 12 months that would limit compliance with study requirements.

Use of herbal products that may decrease PSA levels (e.g., saw palmetto)

Participants who have had cytotoxic chemotherapy for metastatic castration-resistant prostate cancer within the past 3 months. (Participants who have had docetaxel for metastatic castration sensitive per Chemohormonal Therapy Versus Androgen Ablation Randomized Trial for Extensive Disease in Prostate Cancer (CHAARTED) data may enroll as long as they did not have progressive disease while on docetaxel and are 3 months removed from treatment, with all treatment related toxicities resolving to at least grade 1.)

Participants who have undergone major surgery within 4 weeks of enrollment. A biopsy will not preclude a participant from starting study.

Participants with a history of hepatitis B (HBV) are excluded due to potential risk for viral reactivation and resulting liver injury in persons with latent HBV

Subjects unwilling to accept blood products or blood transfusions as medically indicated. As there is a risk of severe bleeding with M7824, participants must be willing to receive blood transfusions if medically necessary for their own safety

For participants enrolling in Arm 2.3A and for participants who may be randomized to Arm 2.3B, the following additional exclusion criteria will apply:

* Subjects receiving Monoamine Oxidase Inhibitors (MAOIs) or a drug which has significant MAOI activity (meperidine, linezolid, methylene blue) within the 21 days before initiation of study therapy are excluded.
* Since epacadostats metabolism may be altered by drugs that inhibit uridine diphosphate (UDP)-glucuronosyltransferase, UGT1A9 (see Appendix D), Participants receiving such drugs within 21 days of initiation of study therapy are excluded.
* Participants receiving agents that are substrates of Cytochrome P450 1A2 (CYP1A2), cytochrome P450 2C8 (CYP2C8), and cytochrome P450 2C19 (CYP2C19) or affected by organic anion transporting polypeptide 1B1 (OATP1B1) or organic anion transporting polypeptide 1B3 (OATP1B3) within 21 days of initiation of study therapy or 5 half-lives of the agent (whichever is shorter) are excluded. Participants receiving medications that are substrates of these enzymes/transporters but are not listed in the appendix or participants receiving substrates of CYP2B6 and CYP3A will be evaluated on a case-by-case basis prior to enrollment. Participants who consume caffeine are eligible but must agree to moderate consumption.
* Subjects receiving coumarin-based anticoagulants (e. Coumadin) are excluded.
* Subjects having any history of Serotonin Syndrome (SS) after receiving serotonergic drugs are excluded.

  --Participants with a QTc corrected for heart rate by Fridericia's formula (QTcF) interval > 480 milliseconds at the screening are excluded. In the event that a single QTcF is > 480 milliseconds, the subject may enroll if the average QTcF for the 3 electrocardiogram (ECG's) is < 480 milliseconds. For subjects with an intraventricular conduction delay (QRS interval > 120 milliseconds), the corrected JT interval, (JTc) interval may be used in place of the QTc. The JTc must be < 340 milliseconds if JTc is used in place of the QTc. QTc prolongation due to pacemaker may enroll if the JTc is normal.
* Subjects with left bundle branch block are excluded.
* Pregnant women are excluded from this study because investigational agents used in this study (BN-Brachyury, M7824, N-803, and/or Epacadostat) could have teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these investigational agents, breastfeeding should be discontinued if the mother is treated with either of them.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James L Gulley, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- [Derived] Fabian KP, Padget MR, Fujii R, Schlom J, Hodge JW. Differential combination immunotherapy requirements for inflamed (warm) tumors versus T cell excluded (cool) tumors: engage, expand, enable, and evolve. J Immunother Cancer. 2021 Feb;9(2):e001691. doi: 10.1136/jitc-2020-001691. PMID 33602696
- [Derived] Redman JM, Steinberg SM, Gulley JL. Quick efficacy seeking trial (QuEST1): a novel combination immunotherapy study designed for rapid clinical signal assessment metastatic castration-resistant prostate cancer. J Immunother Cancer. 2018 Sep 18;6(1):91. doi: 10.1186/s40425-018-0409-8. PMID 30227893
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-C-0078.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase (Ph) I Dose Escalation, Cohort 1, Arm 1.1, Dose Level (DL) 1: Phase I Dose Escalation, Cohort 1, Arm 1.1, Dose Level 1 Participants with any solid tumor M7824 + N-803 (accrual closed) N803 Dose Level 1 =10mcg/kg, M7824 Dose Level 1 =1200mg
- Phase I Dose Escalation, Cohort 1, Arm 1.1 Dose Level 2: Phase I Dose Escalation, Cohort 1, Arm 1.1 Dose Level 2 Participants with any solid tumor M7824 + N-803 (accrual closed) N803 Dose Level 2 = 15mcg/kg M7824 Dose Level 2=1200mg
- Phase I Dose Escalation, Cohort 1: Enrolled But Not Treated: Phase I Dose Escalation, Cohort 1 Participants with any solid tumor M7824 + N-803 (accrual closed)
- Phase IIA Dose Expansion (Dose Exp.), Cohort 2, Arm 2.1A: Phase IIA Dose Expansion, Cohort 2, Arm 2.1A Participants with castration-resistant prostate cancer (CRPC) during Phase IIA M7824 + BN-Brachyury
- Phase IIA Dose Expansion, Cohort 2, Arm 2.2A: Phase IIA Dose Expansion, Cohort 2, Arm 2.2A Participants with CRPC during Phase IIA M7824 + BN-Brachyury + N-803 during phase IIA N803 Dose Level 2 = 15mcg/kg M7824 Dose Level 2=1200mg
- Phase IIB, Dose Expansion, Cohort 2, Arm 2.2B: Phase IIB Dose Expansion, Cohort 2, Arm 2.B Participants with CRPC requiring randomization in phase IIB M7824 + BN-Brachyury during phase IIB + N803 Dose Level 2 = 15mcg/kg M7824 Dose Level 2=1200mg
- Phase IIA Dose Expansion, Cohort 2A, Arm 2.3A: Phase IIA Dose Expansion, Cohort 2A, Arm 2.3A Participants with CRPC during Phase IIA M7824 + BN-Brachyury + N-803 + Epacadostat during phase IIA
Period: Phase I Dose Escalation
Arm/Group | Phase (Ph) I Dose Escalation, Cohort 1, Arm 1.1, Dose Level (DL) 1 | Phase I Dose Escalation, Cohort 1, Arm 1.1 Dose Level 2 | Phase I Dose Escalation, Cohort 1: Enrolled But Not Treated | Phase IIA Dose Expansion (Dose Exp.), Cohort 2, Arm 2.1A | Phase IIA Dose Expansion, Cohort 2, Arm 2.2A | Phase IIB, Dose Expansion, Cohort 2, Arm 2.2B | Phase IIA Dose Expansion, Cohort 2A, Arm 2.3A
Started | 4 | 10 | 1 | 0 | 0 | 0 | 0
Completed | 4 | 9 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Ineligible | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — New therapy | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Phase II Dose Expansion
Arm/Group | Phase (Ph) I Dose Escalation, Cohort 1, Arm 1.1, Dose Level (DL) 1 | Phase I Dose Escalation, Cohort 1, Arm 1.1 Dose Level 2 | Phase I Dose Escalation, Cohort 1: Enrolled But Not Treated | Phase IIA Dose Expansion (Dose Exp.), Cohort 2, Arm 2.1A | Phase IIA Dose Expansion, Cohort 2, Arm 2.2A | Phase IIB, Dose Expansion, Cohort 2, Arm 2.2B | Phase IIA Dose Expansion, Cohort 2A, Arm 2.3A
Started | 4 | 9 | 0 | 13 | 13 | 12 | 6
Follow up Period Completed | 2 | 5 | 0 | 7 | 11 | 7 | 6
Disease Progression on Study | 1 | 2 | 0 | 7 | 8 | 9 | 1
Completed | 4 | 9 | 0 | 10 | 12 | 11 | 6
Not Completed | 0 | 0 | 0 | 3 | 1 | 1 | 0
Not completed — Refused further treatment | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Switched to alternative therapy | 0 | 0 | 0 | 3 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data collected for one participant who was enrolled and not treated is reported here.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase (Ph) I Dose Escalation, Cohort 1, Arm 1.1, Dose Level (DL) 1 | Phase I Dose Escalation, Cohort 1, Arm 1.1 Dose Level 2 | Phase I Dose Escalation, Cohort 1: Enrolled But Not Treated | Phase IIA Dose Expansion (Dose Exp.), Cohort 2, Arm 2.1A | Phase IIA Dose Expansion, Cohort 2, Arm 2.2A | Phase IIB, Dose Expansion, Cohort 2, Arm 2.2B | Phase IIA Dose Expansion, Cohort 2A, Arm 2.3A | Total
Number analyzed (Participants) | 4 | 10 | 1 | 13 | 13 | 12 | 6 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 9 | 1 | 5 | 6 | 6 | 1 | 31
  >=65 years | 1 | 1 | 0 | 8 | 7 | 6 | 5 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.23 (12.56) | 52.34 (12.05) | 50.5 (0) | 67.81 (9.23) | 65.69 (6.81) | 66.57 (6.97) | 75.47 (8.44) | 64.03 (11.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 1 | 0 | 0 | 0 | 0 | 8
  Male | 1 | 6 | 0 | 13 | 13 | 12 | 6 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 1 | 2 | 0 | 0 | 6
  Not Hispanic or Latino | 3 | 7 | 1 | 12 | 9 | 12 | 6 | 50
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 4 | 1 | 5 | 0 | 10
  White | 3 | 9 | 1 | 8 | 8 | 7 | 6 | 42
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 4 | 10 | 1 | 13 | 13 | 12 | 6 | 59

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit With Any of a Set of 3 Possible Treatments for Participants With Metastatic Castration-resistant Prostate Cancer (mCRPC) Reported With an 80% Confidence Interval
Description: Objective clinical response and/or prostate-specific antigen (PSA) decline of >=30% sustained for a minimum of 21 days. Any of these is considered 'clinical benefit.' Objective response was assessed by the response evaluation criteria in solid tumors (RECIST) 1.1. Complete response (CR) is disappearance of all non-target lesions and normalization of tumor marker level. Partial response (PR) is at least a 30% decrease in the sum of the diameters of target lesions. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. Progressive disease (PD) is at least a 20% increase in the sum of the diameters of target lesions. Three treatments evaluated are: Phase II Bavarian Nordic (BN) Brachyury + Bintrafusp alfa (M7824), Phase II Bavarian Nordic (BN) Brachyury + Bintrafusp alfa (M7824) + Anktiva (N-803), and Phase II Bavarian Nordic (BN) Brachyury + Bintrafusp alfa (M7824) + Anktiva (N-803) + Epacadostat.
Time Frame: From enrollment up to 49 weeks
Population: 43/59 participants were analyzed because 14 were not applicable for this endpoint per protocol, 1 was ineligible and 1 was not able to be assessed for this endpoint because participant withdrew from the study before having efficacy assessments.
Measure: Number (80% Confidence Interval); unit: Proportion of participants
Groups:
- All Participants in Phase IIA Dose Expansion and Phase IIB Dose Expansion: Phase IIA Dose Expansion, Cohort 2, Arm 2.2A Participants with CRPC during Phase IIA M7824 + BN-Brachyury + N-803 during phase IIA N803 Dose Level 2 = 15mcg/kg M7824 Dose Level 2=1200mg and Phase IIB Dose Expansion, Cohort 2, Arm 2.B Participants with CRPC requiring randomization in phase IIB M7824 + BN-Brachyury during phase IIB + N803 Dose Level 2 = 15mcg/kg M7824 Dose Level 2=1200mg.
Arm/Group | Phase IIA Dose Expansion (Dose Exp.), Cohort 2, Arm 2.1A | All Participants in Phase IIA Dose Expansion and Phase IIB Dose Expansion | Phase IIA Dose Expansion, Cohort 2A, Arm 2.3A
Number analyzed (Participants) | 13 | 24 | 6
Proportion of participants | .076 [0.0081 to 0.268] | 0.292 [0.170 to 0.442] | 0 [0.000 to 0.319]

2. Primary Outcome: Clinical Benefit(Objective Response if Measurable Disease by Response Evaluation Criteria in Solid Tumors v1.1)With Any of 3 Possible Treatments for Participants With Metastatic Castration-resistant Prostate Cancer Reported With a 95% Confidence Interval
Description: Objective response was assessed by the response evaluation criteria in solid tumors (RECIST) 1.1. Complete response (CR) is disappearance of all non-target lesions and normalization of tumor marker level. Partial response (PR) is at least a 30% decrease in the sum of the diameters of target lesions. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. Progressive disease (PD) is at least a 20% increase in the sum of the diameters of target lesions. Three treatments evaluated are: Phase II Bavarian Nordic (BN) Brachyury + Bintrafusp alfa (M7824), Phase II Bavarian Nordic (BN) Brachyury + Bintrafusp alfa (M7824) + Anktiva (N-803), and Phase II Bavarian Nordic (BN) Brachyury + Bintrafusp alfa (M7824) + Anktiva (N-803) + Epacadostat.
Time Frame: From enrollment up to 49 weeks
Population: 43/59 participants were analyzed because 14 were not applicable for this endpoint per protocol, 1 was ineligible, and 1 was not able to be assessed for this endpoint because participant withdrew from the study before having efficacy assessments.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Phase IIA Dose Expansion (Dose Exp.), Cohort 2, Arm 2.1A | All Participants in Phase IIA Dose Expansion and Phase IIB Dose Expansion | Phase IIA Dose Expansion, Cohort 2A, Arm 2.3A
Number analyzed (Participants) | 13 | 24 | 6
Proportion of participants
  Complete Response | 0 [0.000 to 0.708] | 0 [0.000 to 0.459] | 0 [0.000 to 0.975]
  Partial Response | 0 [0.000 to 0.708] | 0.33 [0.0433 to 0.777] | 0 [0.000 to 0.975]
  Stable Disease | 0.33 [0.0084 to 0.906] | 0 [0.000 to 0.459] | 0 [0.000 to 0.975]
  Progressive Disease | 0.67 [0.0943 to 0.9916] | 0.67 [0.223 to 0.957] | 1 [0.025 to 1.000]

3. Primary Outcome: Phase I/II: Number of Participants With Grades 3, 4, and/or 5 Serious and/or Non-serious Dose-limiting Toxicities (DLT)
Description: A DLT is defined as any of the following adverse events (AE) possibly related to study drugs that occur within 21 days of the start of treatment. Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Grade 3 is moderate. Grade 4 is life-threatening, and Grade 5 is death related to AE. A DLT is any grade ≥ 4 hematologic toxicity or grade 3 thrombocytopenia with associated bleeding; any grade ≥ 3 non-hematologic toxicity, except for any of the following: transient (≤ 48 hour) grade 3 fatigue, local reactions, flu-like symptoms, fever, headache, or nausea, emesis, and diarrhea; or CTCAE Grade 3 skin toxicity lasting less than five days. A non-serious AE is any untoward medical occurrence. A serious AE is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, or congenital anomaly/birth defect.
Time Frame: Within 21 days of the start of treatment
Population: 58/59 participants were analyzed because 1 was ineligible.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase (Ph) I Dose Escalation, Cohort 1, Arm 1.1, Dose Level (DL) 1 | Phase I Dose Escalation, Cohort 1, Arm 1.1 Dose Level 2 | Phase IIA Dose Expansion (Dose Exp.), Cohort 2, Arm 2.1A | Phase IIA Dose Expansion, Cohort 2, Arm 2.2A | Phase IIB, Dose Expansion, Cohort 2, Arm 2.2B | Phase IIA Dose Expansion, Cohort 2A, Arm 2.3A
Number analyzed (Participants) | 4 | 10 | 13 | 13 | 12 | 6
Participants
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: 6-month Progression Free Survival (PFS) Probability
Description: 6-month progression free survival was measured from the on-study date until progression or death without progression in participants and reported with a 95% confidence interval. Progression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The appearance of one or more new lesions is also considered progressions.
Time Frame: 6-months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: proportion probability
Groups:
- All Participants in Phase IIA Dose Expansion and Phase IIB, Dose Expansion: Phase IIA Dose Expansion, Cohort 2, Arm 2.2A. Participants with CRPC during Phase IIA M7824 + BN-Brachyury + N-803 during phase IIA N803 Dose Level 2 = 15mcg/kg M7824 Dose Level 2=1200mg and Phase IIB Dose Expansion, Cohort 2, Arm 2.B. Participants with CRPC requiring randomization in phase IIB M7824 + BN-Brachyury during phase IIB + N803 Dose Level 2 = 15mcg/kg M7824 Dose Level 2=1200mg
Arm/Group | Phase IIA Dose Expansion (Dose Exp.), Cohort 2, Arm 2.1A | Phase IIA Dose Expansion, Cohort 2A, Arm 2.3A | All Participants in Phase IIA Dose Expansion and Phase IIB, Dose Expansion
Number analyzed (Participants) | 13 | 24 | 6
proportion probability | 0.354 [0.152 to 0.822] | 0.348 [0.196 to 0.617] | NA [NA to NA] — Since no participant was followed past 6 months for progression in arm 2.3, the 6-month PFS confidence interval (CI) is not estimable as well.

5. Secondary Outcome: Number of Participants With Grades 1, 2, 3, and 4 Non-serious Adverse Events Related to Treatment Treated With Combinations and Bintrafusp Alfa (M7824) + Anktiva (N-803)
Description: Number of participants with grades 1, 2, 3, and 4 non-serious adverse events related to treatment treated with combinations and Bintrafusp alfa (M7824) + Anktiva (N-803).
Time Frame: 3 weeks dose-limiting toxicity (DLT) period
Measure: Count of Participants; unit: Participants
Arm/Group | Phase (Ph) I Dose Escalation, Cohort 1, Arm 1.1, Dose Level (DL) 1 | Phase I Dose Escalation, Cohort 1, Arm 1.1 Dose Level 2 | Phase IIA Dose Expansion (Dose Exp.), Cohort 2, Arm 2.1A | Phase IIA Dose Expansion, Cohort 2, Arm 2.2A | Phase IIB, Dose Expansion, Cohort 2, Arm 2.2B | Phase IIA Dose Expansion, Cohort 2A, Arm 2.3A
Number analyzed (Participants) | 4 | 10 | 13 | 13 | 12 | 6
Participants
  Grade 1 Anorexia possibly related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 0 | 4 | 0 | 0
  Grade 1 Arthralgia possibly related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Aspartate aminotransferase increased possibly related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Bloating possibly related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Blood and lymphatic system disorders possibly related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Chills possibly related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 0 | 3 | 0 | 0
  Grade 1 Diarrhea possibly related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Dizziness possibly related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 0 | 1 | 0 | 1
  Grade 1 Endocrine disorders - Other specify possibly related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 0 | 2 | 0 | 0
  Grade 1 Fatigue possibly related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 3 | 4 | 0 | 1
  Grade 1 Fever possibly related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 0 | 5 | 0 | 0
  Grade 1 Flatulence possibly related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Flu-like symptoms possibly related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 1 | 6 | 0 | 2
  Grade 1 Headache possibly related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 1 | 1 | 0 | 0
  Grade 1 Hematuria possibly related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Hyperhidrosis possibly related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Injection site reaction possibly related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Insomnia possibly related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 0 | 0 | 0 | 1
  Grade 1 Malaise possibly related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Myalgia possibly related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Nausea possibly related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 1 | 2 | 0 | 0
  Grade 1 Pruritus possibly related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Skin and subcutaneous tissue disorders possibly related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Vertigo possibly related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Vomiting possibly related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Chills probably related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Dizziness probably related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Fatigue probably related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 2 | 0 | 0 | 0
  Grade 1 Fever probably related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 2 | 0 | 0 | 0
  Grade 1 Flu-like symptoms probably related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 2 | 0 | 0 | 0
  Grade 1 Headache probably related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Hyperthyroidism probably related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Injection site reaction probably related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 5 | 0 | 0 | 0
  Grade 1 Malaise probably related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Nausea probably related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 2 | 0 | 0 | 0
  Grade 1 Pain probably related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Chills definitely related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 2 | 0 | 0 | 0
  Grade 1 Fever definitely related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Injection site reaction definitely related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 9 | 7 | 0 | 2
  Grade 1 Pruritus definitely related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Skin and subcutaneous tissue disorders definitely related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 Alanine aminotransferase increased possibly related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 Dehydration possibly related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 Endocrine disorders - Other specify possibly related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 0 | 2 | 0 | 1
  Grade 2 Fatigue possibly related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 1 | 0 | 0 | 1
  Grade 2 Fever possibly related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 Flu-like symptoms possibly related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 Chills probably related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 Hyperhidrosis probably related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 Injection site reaction probably related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 Lipase increased probably related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Injection site reaction definitely related to Bavarian-Nordic (BN)-brachyury | 0 | 0 | 2 | 1 | 0 | 0
  Grade 1 Abdominal pain possibly related to Anktiva (N803) | 0 | 0 | 0 | 0 | 0 | 1
  Grade 1 Anorexia possibly related to Anktiva (N803) | 0 | 0 | 0 | 0 | 0 | 1
  Grade 1 Fatigue possibly related to Anktiva (N803)0 | 0 | 0 | 0 | 0 | 0 | 2
  Grade 1 Insomnia possibly related to Anktiva (N803) | 0 | 0 | 0 | 0 | 0 | 1
  Grade 1 Mucositis oral possibly related to Anktiva (N803) | 0 | 0 | 0 | 0 | 0 | 1
  Grade 1 Pruritus possibly related to Anktiva (N803) | 0 | 0 | 0 | 0 | 0 | 2
  Grade 1 Rash maculo-papular possibly related to Anktiva (N803) | 0 | 0 | 0 | 0 | 0 | 1
  Grade 1 Weight loss possibly related to Anktiva (N803) | 0 | 0 | 0 | 0 | 0 | 1
  Grade 1 Pruritus probably related to Anktiva (N803) | 0 | 0 | 0 | 0 | 0 | 1
  Grade 1 Rash maculo-papular probably related to Anktiva (N803) | 0 | 0 | 0 | 0 | 0 | 4
  Grade 1 Hemoglobinuria definitely related to Anktiva (N803) | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Anorexia possibly related to Anktiva (N803) | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Fatigue possibly related to Anktiva (N803) | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Mucositis oral possibly related to Anktiva (N803) | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Rash maculo-papular possibly related to Anktiva (N803) | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Weight loss possibly related to Anktiva (N803) | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Pruritus probably related to Anktiva (N803) | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Rash maculo-papular probably related to Anktiva (N803) | 0 | 0 | 0 | 0 | 0 | 3
  Grade 3 Rash maculo-papular possibly related to Anktiva (N803) | 0 | 0 | 0 | 0 | 0 | 1
  Grade 3 Pruritus probably related to Anktiva (N803) | 0 | 0 | 0 | 0 | 0 | 1
  Grade 3 Rash maculo-papular probably related to Anktiva (N803) | 0 | 0 | 0 | 0 | 0 | 1
  Grade 1 Abdominal pain possibly related to Epacadostat | 0 | 0 | 0 | 0 | 0 | 1
  Grade 1 Anorexia possibly related to Epacadostat | 0 | 0 | 0 | 0 | 0 | 1
  Grade 1 Fatigue possibly related to Epacadostat | 0 | 0 | 0 | 0 | 0 | 2
  Grade 1 Insomnia possibly related to Epacadostat | 0 | 0 | 0 | 0 | 0 | 1
  Grade 1 Mucositis oral possibly related to Epacadostat | 0 | 0 | 0 | 0 | 0 | 1
  Grade 1 Pruritus possibly related to Epacadostat | 0 | 0 | 0 | 0 | 0 | 2
  Grade 1 Rash maculo-papular possibly related to Epacadostat | 0 | 0 | 0 | 0 | 0 | 1
  Grade 1 Weight loss possibly related to Epacadostat | 0 | 0 | 0 | 0 | 0 | 1
  Grade 1 Pruritus probably related to Epacadostat | 0 | 0 | 0 | 0 | 0 | 1
  Grade 1 Rash maculo-papular probably related to Epacadostat | 0 | 0 | 0 | 0 | 0 | 4
  Grade 1 Hemoglobinuria definitely related to Epacadostat | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Anorexia possibly related to Epacadostat | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Fatigue possibly related to Epacadostat | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Mucositis oral possibly related to Epacadostat | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Weight loss possibly related to Epacadostat | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Pruritus probably related to Epacadostat | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Rash maculo-papular probably related to Epacadostat | 0 | 0 | 0 | 0 | 0 | 3
  Grade 2 Rash maculo-papular possibly related to Epacadostat | 0 | 0 | 0 | 0 | 0 | 1
  Grade 3 Pruritus probably related to Epacadostat | 0 | 0 | 0 | 0 | 0 | 1
  Grade 3 Rash maculo-papular probably related to Epacadostat | 0 | 0 | 0 | 0 | 0 | 1
  Grade 1 Abdominal pain possibly related to M7824 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 1 Alanine aminotransferase increased possibly related to M7824 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Anal hemorrhage possibly related to M7824 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Anorexia possibly related to M7824 | 0 | 2 | 0 | 1 | 0 | 0
  Grade 1 Aspartate aminotransferase increased possibly related to M7824 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Bloating possibly related to M7824 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Blood and lymphatic system disorders - Other specify possibly related to M7824 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Chills possibly related to M7824 | 2 | 1 | 0 | 0 | 0 | 0
  Grade 1 Dry mouth possibly related to M7824 | 0 | 0 | 1 | 2 | 0 | 0
  Grade 1 Dry skin possibly related to M7824 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Endocrine disorders - Other specify possibly related to M7824 | 0 | 0 | 0 | 2 | 0 | 0
  Grade 1 Eosinophilia possibly related to M7824 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Epistaxis possibly related to M7824 | 0 | 1 | 0 | 3 | 0 | 1
  Grade 1 Eye disorders - Other specify possibly related to M7824 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Fatigue possibly related to M7824 | 1 | 3 | 6 | 3 | 0 | 0
  Grade 1 Fever possibly related to M7824 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 1 Flatulence possibly related to M7824 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Flu-like symptoms possibly related to M7824 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Gastrointestinal disorders - Other specify possibly related to M7824 | 0 | 0 | 3 | 2 | 0 | 0
  Grade 1 Generalized muscle weakness possibly related to M7824 | 1 | 0 | 0 | 0 | 0 | 0
  Grade 1 Headache possibly related to M7824 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 1 Hematuria possibly related to M7824 | 0 | 1 | 3 | 1 | 0 | 1
  Grade 1 Hemolysis possibly related to M7824 | 0 | 1 | 0 | 0 | 0 | 1
  Grade 1 Hemorrhoidal hemorrhage possibly related to M7824 | 0 | 0 | 1 | 1 | 0 | 0
  Grade 1 Hoarseness possibly related to M7824 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Hypothyroidism possibly related to M7824 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Insomnia possibly related to M7824 | 0 | 0 | 0 | 0 | 0 | 1
  Grade 1 Malaise possibly related to M7824 | 0 | 1 | 1 | 0 | 0 | 0
  Grade 1 Mucositis oral possibly related to M7824 | 0 | 0 | 0 | 0 | 0 | 1
  Grade 1 Nausea possibly related to M7824 | 0 | 2 | 1 | 0 | 0 | 0
  Grade 1 Pain possibly related to M7824 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 1 Pruritus possibly related to M7824 | 0 | 2 | 0 | 3 | 0 | 2
  Grade 1 Rash maculo-papular possibly related to M7824 | 0 | 1 | 2 | 3 | 0 | 1
  Grade 1 Sinus tachycardia possibly related to M7824 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Skin and subcutaneous tissue disorders - Other specify possibly related to M7824 | 0 | 1 | 1 | 1 | 0 | 0
  Grade 1 Thyroid stimulating hormone possibly related to M7824 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 1 Alanine aminotransferase increased probably related to M7824 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Alkaline phosphatase increased probably related to M7824 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Aspartate aminotransferase increased probably related to M7824 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Cystitis noninfective probably related to M7824 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Dry skin probably related to M7824 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Endocrine disorders - Other specify probably related to M7824 | 0 | 0 | 1 | 1 | 0 | 0
  Grade 1 Enterocolitis probably related to M7824 | 0 | 2 | 0 | 0 | 0 | 0
  Grade 1 Eosinophilia probably related to M7824 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Fatigue probably related to M7824 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Gastrointestinal disorders - Other specify probably related to M7824 | 0 | 0 | 0 | 0 | 0 | 1
  Grade 1 General disorders and administration site conditions probably related to M7824 | 0 | 0 | 0 | 2 | 0 | 0
  Grade 1 Gingival pain probably related to M7824 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 1 Hematuria probably related to M7824 | 0 | 0 | 1 | 1 | 0 | 0
  Grade 1 Hyperthyroidism probably related to M7824 | 0 | 0 | 1 | 1 | 0 | 1
  Grade 1 Hypotension probably related to M7824 | 1 | 0 | 0 | 0 | 0 | 0
  Grade 1 Hypothyroidism probably related to M7824 | 0 | 0 | 0 | 1 | 0 | 1
  Grade 1 Lipase increased probably related to M7824 | 0 | 0 | 0 | 3 | 0 | 1
  Grade 1 Metabolism and nutrition disorders - Other specify probably related to M7824 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Neoplasms benign, malignant and unspecified incl cysts and polyps probably related to M7824 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 1 Oral hemorrhage probably related to M7824 | 0 | 0 | 2 | 0 | 0 | 1
  Grade 1 Pruritus probably related to M7824 | 0 | 0 | 1 | 1 | 0 | 0
  Grade 1 Rash acneiform probably related to M7824 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 1 Rash maculo-papular probably related to M7824 | 1 | 3 | 0 | 5 | 0 | 0
  Grade 1 Serum amylase probably related to M7824 | 0 | 0 | 0 | 2 | 0 | 0
  Grade 1 Skin and subcutaneous tissue disorders - Other specify probably related to M7824 | 0 | 0 | 1 | 1 | 0 | 0
  Grade 1 Thyroid stimulating hormone increased probably related to M7824 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 1 Bullous dermatitis definitely related to M7824 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 1 Hyperkeratosis definitely related to M7824 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Hypothyroidism definitely related to M7824 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Infusion related reaction definitely related to M7824 | 1 | 0 | 0 | 1 | 0 | 0
  Grade 1 Injection site reaction definitely related to M7824 | 0 | 2 | 0 | 0 | 0 | 0
  Grade 1 Paresthesia definitely related to M7824 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Periorbital edema probably related to M7824 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Skin and subcutaneous tissue disorders - Other specify definitely related to M7824 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 Alanine aminotransferase increased possibly related to M7824 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 Anal hemorrhage possibly related to M7824 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 Anemia possibly related to M7824 | 0 | 2 | 0 | 1 | 0 | 1
  Grade 2 Diarrhea possibly related to M7824 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 Dry mouth possibly related to M7824 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 Endocrine disorders - Other specify possibly related to M7824 | 0 | 0 | 0 | 2 | 0 | 1
  Grade 2 Eye disorders possibly related to M7824 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 Fatigue possibly related to M7824 | 0 | 3 | 1 | 1 | 0 | 0
  Grade 2 Fever possibly related to M7824 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 General disorders and administration site conditions-Other specify possibly related to M7824 | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Hematuria possibly related to M7824 | 0 | 0 | 0 | 1 | 0 | 2
  Grade 2 Hypotension possibly related to M7824 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 Joint range of motion decreased possibly related to M7824 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 Lipase increased possibly related to M7824 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 Lymphocyte count decreased possibly related to M7824 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 Mucositis oral possibly related to M7824 | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Musculoskeletal and connective tissue disorder Other specify possibly related to M7824 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 Nausea possibly related to M7824 | 1 | 0 | 0 | 0 | 0 | 0
  Grade 2 Pain possibly related to M7824 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 Proteinuria possibly related to M7824 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 Pruritus possibly related to M7824 | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Rash maculo-papular possibly related to M7824 | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Skin and subcutaneous tissue disorders Other specify possibly related to M7824 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 Small intestine ulcer possibly related to M7824 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 Vomiting possibly related to M7824 | 2 | 0 | 0 | 0 | 0 | 0
  Grade 2 Anemia probably related to M7824 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 Bullous dermatitis probably related to M7824 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 Dry mouth probably related to M7824 | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Endocrine disorders - Other specify probably related to M7824 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 Eye disorders probably related to M7824 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 Hyperthyroidism probably related to M7824 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 Hypothyroidism probably related to M7824 | 0 | 1 | 1 | 2 | 0 | 0
  Grade 2 Infusion related reaction probably related to M7824 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 Lipase increased probably related to M7824 | 0 | 0 | 0 | 4 | 0 | 1
  Grade 2 Proctitis probably related to M7824 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 Rash maculo-papular probably related to M7824 | 0 | 1 | 0 | 2 | 0 | 0
  Grade 2 Serum amylase probably related to M7824 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 Skin and subcutaneous tissue disorders - Other specify probably related to M7824 | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Urticaria probably related to M7824 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 Arthritis definitely related to M7824 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 Infusion related reaction definitely related to M7824 | 0 | 0 | 0 | 1 | 0 | 2
  Grade 2 Pruritus definitely related to M7824 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 Skin and subcutaneous tissue disorders Other specify definitely related to M7824 | 0 | 0 | 0 | 0 | 0 | 1
  Grade 3 Anemia possibly related to M7824 | 0 | 0 | 0 | 0 | 0 | 1
  Grade 3 Blood and lymphatic system disorders Other specify possibly related to M7824 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 Gastrointestinal disorders Other specify possibly related to M7824 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 3 Rash maculopapular possibly related to M7824 | 0 | 0 | 0 | 0 | 0 | 1
  Grade 3 Eosinophilia probably related to M7824 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 Lipase increased probably related to M7824 | 0 | 0 | 0 | 0 | 0 | 1
  Grade 3 Pancreatitis probably related to M7824 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Alanine aminotransferase increased possibly related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Aspartate aminotransferase increased possibly related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Dizziness possibly related to research | 0 | 0 | 0 | 1 | 0 | 1
  Grade 1 Dry skin possibly related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Endocrine disorders Other specify possibly related to research | 0 | 0 | 0 | 2 | 0 | 0
  Grade 1 Eosinophilia possibly related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Eye disorders Other specify possibly related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Fever possibly related to research | 0 | 0 | 0 | 5 | 0 | 0
  Grade 1 Hemolysis possibly related to research | 0 | 0 | 0 | 0 | 0 | 1
  Grade 1 Hyperhidrosis possibly related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Injection site reaction possibly related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Insomnia possibly related to research | 0 | 0 | 0 | 0 | 0 | 1
  Grade 1 Malaise possibly related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Mucositis oral possibly related to research | 0 | 0 | 0 | 0 | 0 | 1
  Grade 1 Myalgia possibly related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Vertigo possibly related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Weight loss possibly related to research | 0 | 0 | 0 | 0 | 0 | 1
  Grade 1 Anal hemorrhage possibly related to research | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Arthralgia possibly related to research | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Bloating possibly related to research | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Blood and lymphatic system disorders Other specify possibly related to research | 0 | 0 | 1 | 1 | 0 | 0
  Grade 1 Diarrhea possibly related to research | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Dry mouth possibly related to research | 0 | 0 | 1 | 2 | 0 | 0
  Grade 1 Flatulence possibly related to research | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Flu-like symptoms possibly related to research | 0 | 0 | 1 | 6 | 0 | 2
  Grade 1 Hemorrhoidal hemorrhage possibly related to research | 0 | 0 | 1 | 1 | 0 | 0
  Grade 1 Hoarseness possibly related to research | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Hypothyroidism possibly related to research | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Sinus tachycardia possibly related to research | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Vomiting possibly related to research | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Pain possibly related to research | 0 | 1 | 0 | 0 | 0 | 0
  Grade 1 Thyroid stimulating hormone possibly related to research | 0 | 1 | 0 | 0 | 0 | 0
  Grade 1 Alanine aminotransferase increased probably related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Alkaline phosphatase increased probably related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Aspartate aminotransferase increased probably related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Eosinophilia probably related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Gastrointestinal disorders Other specify probably related to research | 0 | 0 | 0 | 0 | 0 | 1
  Grade 1 Hypothyroidism probably related to research | 0 | 0 | 0 | 1 | 0 | 1
  Grade 1 Lipase increased probably related to research | 0 | 0 | 0 | 3 | 0 | 1
  Grade 1 Metabolism and nutrition disorders Other specify probably related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Periorbital edema probably related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Serum amylase probably related to research | 0 | 0 | 0 | 2 | 0 | 0
  Grade 1 Cystitis noninfective probably related to research | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Dry skin probably related to research | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Endocrine disorders Other specify probably related to research | 0 | 0 | 1 | 1 | 0 | 0
  Grade 1 Hematuria probably related to research | 0 | 0 | 1 | 1 | 0 | 0
  Grade 1 Oral hemorrhage probably related to research | 0 | 0 | 2 | 0 | 0 | 1
  Grade 1 Gastrointestinal disorders Other specify possibly related to research | 0 | 0 | 3 | 2 | 0 | 0
  Grade 1 Abdominal pain possibly related to research | 0 | 1 | 0 | 0 | 0 | 1
  Grade 1 Epistaxis possibly related to research | 0 | 1 | 0 | 3 | 0 | 1
  Grade 1 Anorexia possibly related to research | 0 | 1 | 0 | 5 | 0 | 1
  Grade 1 Diarrhea probably related to research | 0 | 1 | 0 | 0 | 0 | 0
  Grade 1 General disorders& administration site conditions Other specify probably related to research | 0 | 1 | 0 | 2 | 0 | 0
  Grade 1 Generalized edema probably related to research | 0 | 1 | 0 | 0 | 0 | 0
  Grade 1 Gingival pain probably related to research | 0 | 1 | 0 | 0 | 0 | 0
  Grade 1 Hyperhidrosis probably related to research | 0 | 1 | 0 | 0 | 0 | 0
  Grade 1 Myalgia probably related to research | 0 | 1 | 0 | 0 | 0 | 0
  Grade 1 Neoplasms benign, malignant and unspecified Other specify probably related to research | 0 | 1 | 0 | 0 | 0 | 0
  Grade 1 Rash acneiform probably related to research | 0 | 1 | 0 | 0 | 0 | 0
  Grade 1 Thyroid stimulating hormone probably related to research | 0 | 1 | 0 | 0 | 0 | 0
  Grade 1 Vomiting probably related to research | 0 | 1 | 0 | 0 | 0 | 0
  Grade 1 Malaise probably related to research | 0 | 1 | 1 | 0 | 0 | 0
  Grade 1 Enterocolitis probably related to research | 0 | 2 | 0 | 0 | 0 | 0
  Grade 1 Anorexia probably related to research | 0 | 3 | 0 | 0 | 0 | 1
  Grade 1 Headache probably related to research | 0 | 3 | 1 | 0 | 0 | 0
  Grade 1 Nausea probably related to research | 0 | 3 | 2 | 1 | 0 | 0
  Grade 1 Fatigue possibly related to research | 0 | 3 | 4 | 3 | 0 | 2
  Grade 1 Chills possibly related to research | 1 | 0 | 0 | 3 | 0 | 0
  Grade 1 Generalized muscle weakness possibly related to research | 1 | 0 | 0 | 0 | 0 | 0
  Grade 1 Dizziness probably related to research | 1 | 0 | 1 | 0 | 0 | 0
  Grade 1 Pain probably related to research | 1 | 0 | 1 | 0 | 0 | 0
  Grade 1 Skin and subcutaneous tissue disorders Other specify probably related to research | 1 | 0 | 1 | 1 | 0 | 0
  Grade 1 Fatigue probably related to research | 1 | 0 | 2 | 1 | 0 | 0
  Grade 1 Flu-like symptoms probably related to research | 1 | 2 | 2 | 2 | 0 | 0
  Grade 1 Rash maculo-papular probably related to research | 1 | 3 | 0 | 5 | 0 | 4
  Grade 1 Injection site reaction probably related to research | 1 | 7 | 5 | 2 | 0 | 0
  Grade 1 Hypotension probably related to research | 2 | 0 | 0 | 0 | 0 | 0
  Grade 1 Pruritus probably related to research | 2 | 1 | 1 | 2 | 0 | 1
  Grade 1 Fever probably related to research | 2 | 5 | 2 | 0 | 0 | 0
  Grade 1 Chills probably related to research | 3 | 8 | 1 | 0 | 0 | 0
  Grade 1 Hyperthyroidism probably related to research | 0 | 0 | 1 | 2 | 0 | 1
  Grade 1 Flu-like symptoms definitely related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Hemoglobinuria definitely related to research | 0 | 0 | 0 | 0 | 0 | 1
  Grade 1 Hypothyroidism definitely related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Paresthesia definitely related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 1 Hyperkeratosis definitely related to research | 0 | 0 | 1 | 0 | 0 | 0
  Grade 1 Skin and subcutaneous tissue disorders Other specify definitely related to research | 0 | 0 | 2 | 0 | 0 | 0
  Grade 1 Bullous dermatitis definitely related to research | 0 | 1 | 0 | 0 | 0 | 0
  Grade 1 Hemolysis definitely related to research | 0 | 1 | 0 | 0 | 0 | 0
  Grade 1 Fever definitely related to research | 0 | 1 | 1 | 1 | 0 | 0
  Grade 1 Nausea possibly related to research | 0 | 1 | 1 | 3 | 0 | 0
  Grade 1 Headache possibly related to research | 0 | 1 | 1 | 1 | 0 | 0
  Grade 1 Skin and subcutaneous tissue disorders Other specify possibly related to research | 0 | 1 | 1 | 1 | 0 | 0
  Grade 1 Rash maculo-papular possibly related to research | 0 | 1 | 2 | 3 | 0 | 1
  Grade 1 Hematuria possibly related to research | 0 | 1 | 3 | 1 | 0 | 1
  Grade 1 Pruritus possibly related to research | 0 | 2 | 0 | 2 | 0 | 2
  Grade 1 Chills definitely related to research | 0 | 2 | 2 | 0 | 0 | 0
  Grade 1 Infusion related reaction definitely related to research | 1 | 0 | 0 | 1 | 0 | 0
  Grade 1 Edema limbs definitely related to research | 1 | 0 | 0 | 0 | 0 | 0
  Grade 1 Skin induration definitely related to research | 1 | 0 | 0 | 0 | 0 | 0
  Grade 1 Pain definitely related to research | 1 | 0 | 0 | 0 | 0 | 0
  Grade 1 Pruritus definitely related to research | 1 | 0 | 1 | 1 | 0 | 0
  Grade 1 Injection site reaction definitely related to research | 4 | 9 | 9 | 10 | 0 | 6
  Grade 2 Weight loss possibly related to research | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Alanine aminotransferase increased possibly related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 Anorexia possibly related to research | 0 | 0 | 0 | 0 | 0 | 1
  Grade 1 Dehydration possibly related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 Endocrine disorders - Other specify possibly related to research | 0 | 0 | 0 | 1 | 0 | 1
  Grade 2 Eye disorders Other specify possibly related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 Hypotension possibly related to research | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 Lipase increased possibly related to research | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 Anal hemorrhage possibly related to research | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 Diarrhea possibly related to research | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 Headache possibly related to research | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 Neutrophil count decreased | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 Pain possibly related to research | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 Proteinuria possibly related to research | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 Sinusitis possibly related to research | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 Fatigue possibly related to research | 0 | 1 | 1 | 1 | 0 | 1
  Grade 2 Lymphocyte count decreased possibly related to research | 0 | 3 | 0 | 0 | 0 | 0
  Grade 2 Anemia possibly related to research | 0 | 3 | 0 | 1 | 0 | 1
  Grade 2 Alkaline phosphatase increased possibly related to research | 1 | 0 | 0 | 0 | 0 | 0
  Grade 2 Vomiting possibly related to research | 2 | 0 | 0 | 0 | 0 | 0
  Grade 2 Nausea possibly related to research | 2 | 0 | 0 | 0 | 0 | 0
  Grade 2 Eye disorders Other specify probably related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 Fever possibly related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 Flu-like symptoms possibly related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 General disorders& administration site conditions Other specify possibly related to research | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Hematuria possibly related to research | 0 | 0 | 0 | 1 | 0 | 2
  Grade 2 Joint range of motion decreased possibly related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 Mucositis oral possibly related to research | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Musculoskeletal and connective tissue disorder Other specify possibly related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 Rash maculo-papular possibly related to research | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Skin and subcutaneous tissue disorders Other specify possibly related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 Hyperthyroidism probably related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 Lipase increased probably related to research | 0 | 0 | 0 | 4 | 0 | 1
  Grade 2 Pruritus probably related to research | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Serum amylase probably related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 Skin and subcutaneous tissue disorders Other, specify, probably related to research | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Urticaria probably related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 Dry mouth probably related to research | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Endocrine disorders other specify probably related to research | 0 | 0 | 0 | 2 | 0 | 0
  Grade 2 Hematuria probably related to research | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 Chills probably related to research | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 Infusion related reaction probably related to research | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 Proctitis probably related to research | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 Hyperhidrosis probably related to research | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 Anemia probably related to research | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 Bullous dermatitis probably related to research | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 Dehydration probably related to research | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 Hyponatremia probably related to research | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 Nausea probably related to research | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 Rash maculo-papular probably related to research | 0 | 1 | 0 | 2 | 0 | 3
  Grade 2 Hypothyroidism probably related to research | 0 | 1 | 1 | 2 | 0 | 0
  Grade 2 Injection site reaction probably related to research | 0 | 1 | 1 | 1 | 0 | 1
  Grade 2 Fatigue probably related to research | 0 | 2 | 0 | 0 | 0 | 0
  Grade 2 Fever probably related to research | 1 | 1 | 0 | 0 | 0 | 0
  Grade 2 Infusion related reaction definitely related to research | 0 | 0 | 0 | 1 | 0 | 2
  Grade 2 Skin and subcutaneous tissue disorders Other specify definitely related to research | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Arthritis definitely related to research | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 Injection site reaction definitely related to research | 0 | 2 | 3 | 7 | 0 | 3
  Grade 2 Pruritus definitely related to research | 1 | 2 | 0 | 0 | 0 | 0
  Grade 3 Anemia possibly related to research | 0 | 0 | 0 | 0 | 0 | 1
  Grade 3 Blood and lymphatic system disorders Other specify possibly related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 Gastrointestinal disorders possibly related to research | 0 | 0 | 1 | 0 | 0 | 0
  Grade 3 Eosinophilia probably related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 Lipase increased probably related to research | 0 | 0 | 0 | 0 | 0 | 1
  Grade 3 Pruritus probably related to research | 0 | 0 | 0 | 0 | 0 | 1
  Grade 3 Rash maculo-papular possibly related to research | 0 | 0 | 0 | 0 | 0 | 1
  Grade 3 Rash maculo-papular probably related to research | 0 | 0 | 0 | 0 | 0 | 1
  Grade 3 Pancreatitis probably related to research | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 Small intestine ulcer possibly related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 injection site reaction definitely related to M7824 | 0 | 0 | 1 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Grades 3, 4, and/or 5 Serious Adverse Events Related to Treatment Treated With Combinations and Bintrafusp Alfa (M7824) + Anktiva (N-803)
Description: Number of participants with grades 3 4, and/or 5 serious adverse events related to treatment treated with combinations and Bintrafusp alfa (M7824) + Anktiva (N-803).
Time Frame: 3 weeks dose-limiting toxicity (DLT) period
Measure: Count of Participants; unit: Participants
Arm/Group | Phase (Ph) I Dose Escalation, Cohort 1, Arm 1.1, Dose Level (DL) 1 | Phase I Dose Escalation, Cohort 1, Arm 1.1 Dose Level 2 | Phase IIA Dose Expansion (Dose Exp.), Cohort 2, Arm 2.1A | Phase IIA Dose Expansion, Cohort 2, Arm 2.2A | Phase IIB, Dose Expansion, Cohort 2, Arm 2.2B | Phase IIA Dose Expansion, Cohort 2A, Arm 2.3A
Number analyzed (Participants) | 4 | 10 | 13 | 13 | 12 | 6
Participants
  Grade 3 Metabolism and nutrition disorders - Other, specify possibly related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 Metabolism and nutrition disorders - Other, specify possibly related to M7824 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 Tumor hemorrhage possibly related to research | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 Tumor hemorrhage possibly related to M7824 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 Endocrine disorders - Other specify probably related to research | 0 | 0 | 1 | 0 | 0 | 0
  Grade 3 Endocrine disorders - Other specify probably related to M7824 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 3 Enterocolitis probably related to research | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 Enterocolitis probably related to M7824 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 Tumor hemorrhage probably related to research | 0 | 0 | 1 | 0 | 0 | 0
  Grade 3 Tumor hemorrhage probably related to M7824 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 4 Blood and lymphatic system disorders - Other specify possibly related to research | 0 | 0 | 0 | 1 | 0 | 0
  Grade 4 Blood and lymphatic system disorders - Other specify possibly related to M7824 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 4 Blood and lymphatic system disorders - Other specify possibly related to Anktiva (N-803) | 0 | 0 | 0 | 1 | 0 | 0
  Grade 5 related to research and/or any study treatment | 0 | 0 | 0 | 0 | 0 | 0

7. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Adverse Events were monitored/assessed from the first study intervention, up to 49 weeks.
Population: 58/59 participants were analyzed because one was deemed ineligible.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase (Ph) I Dose Escalation, Cohort 1, Arm 1.1, Dose Level (DL) 1 | Phase I Dose Escalation, Cohort 1, Arm 1.1 Dose Level 2 | Phase IIA Dose Expansion (Dose Exp.), Cohort 2, Arm 2.1A | Phase IIA Dose Expansion, Cohort 2, Arm 2.2A | Phase IIB, Dose Expansion, Cohort 2, Arm 2.2B | Phase IIA Dose Expansion, Cohort 2A, Arm 2.3A
Number analyzed (Participants) | 4 | 10 | 13 | 13 | 12 | 6
Participants | 4 | 10 | 13 | 13 | 12 | 6

ADVERSE EVENTS:
Time Frame: Adverse Events were monitored/assessed from the first study intervention, up to 49 weeks.
Description: 58/59 participants were analyzed because one was deemed ineligible.
Arm/Group | Phase (Ph) I Dose Escalation, Cohort 1, Arm 1.1, Dose Level (DL) 1 | Phase I Dose Escalation, Cohort 1, Arm 1.1 Dose Level 2 | Phase IIA Dose Expansion (Dose Exp.), Cohort 2, Arm 2.1A | Phase IIA Dose Expansion, Cohort 2, Arm 2.2A | Phase IIB, Dose Expansion, Cohort 2, Arm 2.2B | Phase IIA Dose Expansion, Cohort 2A, Arm 2.3A
All-Cause Mortality (participants affected / at risk) | 1/4 | 2/10 | 1/13 | 0/13 | 0/12 | 0/6
Serious Adverse Events (participants affected / at risk) | 3/4 | 5/10 | 8/13 | 5/13 | 3/12 | 2/6
Other Adverse Events (participants affected / at risk) | 4/4 | 10/10 | 13/13 | 13/13 | 12/12 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase (Ph) I Dose Escalation, Cohort 1, Arm 1.1, Dose Level (DL) 1 (N=4) | Phase I Dose Escalation, Cohort 1, Arm 1.1 Dose Level 2 (N=10) | Phase IIA Dose Expansion (Dose Exp.), Cohort 2, Arm 2.1A (N=13) | Phase IIA Dose Expansion, Cohort 2, Arm 2.2A (N=13) | Phase IIB, Dose Expansion, Cohort 2, Arm 2.2B (N=12) | Phase IIA Dose Expansion, Cohort 2A, Arm 2.3A (N=6)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylaxis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteremia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, specify: Immune mediated neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify: Non-ST elevation myocardial infarction, Type II (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocrine disorders - Other, specify: Isolated ACTH Insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial muscle weakness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify: colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, specify: Mucosal bleeding (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalized edema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify: Human ehrlichiosis and human anaplasmosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify: Infected psoas hematoma (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify: Peritonsillar Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, specify: Immune mediated diabetes (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, specify: Metastasectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase (Ph) I Dose Escalation, Cohort 1, Arm 1.1, Dose Level (DL) 1 (N=4) | Phase I Dose Escalation, Cohort 1, Arm 1.1 Dose Level 2 (N=10) | Phase IIA Dose Expansion (Dose Exp.), Cohort 2, Arm 2.1A (N=13) | Phase IIA Dose Expansion, Cohort 2, Arm 2.2A (N=13) | Phase IIB, Dose Expansion, Cohort 2, Arm 2.2B (N=12) | Phase IIA Dose Expansion, Cohort 2A, Arm 2.3A (N=6)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 4 (7) | 5 (5) | 2 (2) | 1 (2) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 2 (2) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 2 (2) | 1 (1) | 4 (7) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anaphylaxis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (4) | 9 (32) | 3 (7) | 4 (14) | 4 (5) | 2 (5)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 5 (5) | 1 (1) | 8 (13) | 5 (6) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 3 (3) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, specify: Elevated D-Dimer (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood and lymphatic system disorders - Other, specify: Elevated PTT (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood and lymphatic system disorders - Other, specify: Immune-mediated neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, specify: right neck LN (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (6) | 2 (2) | 2 (3)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CPK increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify: Aortic aneurysm (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac disorders - Other, specify: CAD (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify: Coronary Calcification (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 3 (6) | 9 (23) | 3 (4) | 4 (8) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 1 (2) | 3 (5) | 2 (2) | 4 (4) | 3 (4)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Ear and labyrinth disorders - Other, specify: Foreign Body Sensation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema face (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endocrine disorders - Other, specify: Elevated A1C (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endocrine disorders - Other, specify: Isolated ACTH Deficiency (Central AI) (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endocrine disorders - Other, specify: Isolated ACTH Insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (6) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 5 (10) | 1 (1) | 1 (1)
Eye disorders - Other, specify: Double Vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, specify: Iritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Eye disorders - Other, specify: Kaleidoscope vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, specify: L 4th nerve palsy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, specify: Ocular Hypertension (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, specify: Popped blood vessel in right eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, specify: Stye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, specify: Subconjunctival Hemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Facial muscle weakness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 5 (6) | 7 (10) | 8 (25) | 7 (8) | 2 (3)
Fever (General disorders) | 2 (5) | 7 (21) | 3 (6) | 6 (14) | 0 (0) | 0 (0)
Fibrinogen decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 1 (1) | 2 (3) | 4 (6) | 9 (33) | 8 (16) | 3 (3)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
GGT increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, specify: Dilation of pancreatic duct (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify: Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify: Gingival hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify: Hematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (7) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify: colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify: L Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify: Loose stools (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify: Loose stools 2-3/day (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify: Melena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify: hematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify: Groin edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify: Lightheadedness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, specify: Mucosal bleed, blood in urine (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, specify: Phantom Phantosmia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — : Substernal and epigastric pain/discomfort
General disorders and administration site conditions - Other, specify: (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — disease progression, MRI hip and lumbar spine, acetaminophen, radiation
General disorders and administration site conditions - Other, specify: gum bleeding (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 3 (3) | 0 (0)
Generalized edema (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 8 (8) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary disorders - Other, specify: Transaminitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (2) | 3 (5) | 1 (1) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (4) | 0 (0) | 2 (4) | 1 (1) | 1 (1) | 2 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (6) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, specify: Aphthous Ulcer (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 2 (2)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 4 (8) | 10 (85) | 11 (68) | 13 (126) | 12 (32) | 6 (23)
Injury, poisoning and procedural complications - Other, specify: Inguinal hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — : Trauma (Bruise to L cheek from fall at home)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Investigations - Other, specify: Decreased TSH (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Investigations - Other, specify: Elevated Acid Phosphatase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Investigations - Other, specify: Elevated Ferritin (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Investigations - Other, specify: Low iron (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Investigations - Other, specify: Oral plaque-back of throat (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Investigations - Other, specify: TSH Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Joint range of motion decreased lumbar spine (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 6 (16) | 3 (4) | 2 (4)
Localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Lymphedema (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 4 (4) | 2 (5) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, specify: Hypoglycemic Symptoms (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, specify: Immune mediated diabetes (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (2)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify: Anterolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — : Bilateral fingers/hand swelling and stiffness
Musculoskeletal and connective tissue disorder - Other, specify: Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify: Compression fracture L2/L3 (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify: Left fifth digit nodule (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify: Right Hip Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify: Spinal canal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify: Synovitis L ankle (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — : Trigger finger R hand Rand middle finger; L hand ringer
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (5) | 3 (3) | 4 (7) | 5 (8) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — : Brain Metastasis
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — : Cutaneous Squamous Cell Carcinoma
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify: Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — : Keratocanthomas
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (2)
Pain (General disorders) | 1 (3) | 4 (10) | 9 (16) | 7 (10) | 1 (1) | 3 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periorbital edema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (4) | 1 (1) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 3 (4) | 2 (3) | 1 (1) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (6) | 4 (6) | 3 (3) | 6 (11) | 0 (0) | 4 (8)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (8) | 2 (2) | 6 (16) | 2 (2) | 5 (12)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Renal and urinary disorders - Other, specify: B/l hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify: Bladder wall thickening (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify: Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify: Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, specify: Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify: Urinary hesitancy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Reproductive system and breast disorders - Other, specify: Bilateral hydrocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Reproductive system and breast disorders - Other, specify: Left testicular swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify: Influenza (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Serum amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 4 (7) | 2 (2) | 0 (0)
Shingles (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify: Abdominal rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify: Calcinosis cutis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify: Dermatitis Herpetiformis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify: Diaphoresis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify: Keratoacanthoma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify: Keratoacanthoma - R scalp (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify: Keratoacanthoma hand lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify: Keratoacanthomas (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify: Keratoacanthoma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify: Keratoacanthomas (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify: L gluteal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify: Lichenoid dermatitis. (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify: Rash (facial) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — : Rash- contact dermatitis, R & L upper arms, b/l thigh
Skin and subcutaneous tissue disorders - Other, specify: Red spot beneath L nipple (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify: Skin tear, gluteal fold (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Small intestine ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, specify: Biopsy finger, L. third distal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, specify: Left Knee (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, specify: MOHS - Dorsal R hand for SCC and skin graft (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, specify: Oral Surgery - Removal of Surgical Bone (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, specify: Right Craniotomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, specify: Slit his L index finger on home project (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Thrush (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroid stimulating hormone increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular disorders - Other, specify: Cervical Lymphadenopathy (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular disorders - Other, specify: Facial sweating (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Vulval infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight gain (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-17): https://cdn.clinicaltrials.gov/large-docs/45/NCT03493945/Prot_SAP_000.pdf
  • Informed Consent Form (2024-06-25): https://cdn.clinicaltrials.gov/large-docs/45/NCT03493945/ICF_001.pdf